CLINICAL TRIAL: NCT03225950
Title: Interaction Between Immune Cells and Bacteria Associated With Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Anne Katrine Danielsen, Research Assistant, University of Copenhagen
Other Study IDs: H-16024734
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2018-10

CONDITIONS: Periodontal Diseases; Periodontitis; Aggressive Periodontitis; Immunologic Disease; Microbial Disease; Periodontal Pocket; Inflammation; Inflammation Gum; Dysbiosis; Rheumatoid Arthritis; Generalized Aggressive Periodontitis; Generalized Chronic Periodontitis; Chronic Periodontitis
Keywords: Periodontal disease; Periodontitis; Aggressive periodontitis; Dysbiosis; Inflammation; Regulation; Cytokines; Bacteria; Porphyromonas gingivalis; Saliva; Anti-CCP; Peptidyl arginine deiminases; Single nucleotide polymorphisms
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Aggressive Periodontitis; Immune System Diseases; Periodontal Pocket; Inflammation; Gingivitis; Dysbiosis; Arthritis, Rheumatoid; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva, whole blood, peripheral mononuclear blood cells, serum, plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic periodontitis donors: * Donors are medically healthy.
  * Slow to moderate attachment loss and bone destruction.
  * Good correlation between etiological factors and serverity of attachment loss.
  Interventions: Other: In vitro stimulation of blood with periodontitis-associated- and control bacteria; Diagnostic Test: Anti-CCP- and anti-P.g.-antibodies titers; Genetic: Analysis of selected single nucleotide polymorphisms (SNPs); Diagnostic Test: periodontitis-associated bacteria presence
- Aggressive periodontitis donors: * Donors are medically healthy.
  * Rapid attachment loss and bone destruction.
  * Familial aggregation.
  * No correlation between etiological factors and serverity of attachment loss.
  Interventions: Other: In vitro stimulation of blood with periodontitis-associated- and control bacteria; Diagnostic Test: Anti-CCP- and anti-P.g.-antibodies titers; Genetic: Analysis of selected single nucleotide polymorphisms (SNPs); Diagnostic Test: periodontitis-associated bacteria presence
- Control donors: * Donors are medically healthy.
  * No sign of inflammatory conditions.
  Interventions: Other: In vitro stimulation of blood with periodontitis-associated- and control bacteria; Diagnostic Test: Anti-CCP- and anti-P.g.-antibodies titers; Genetic: Analysis of selected single nucleotide polymorphisms (SNPs); Diagnostic Test: periodontitis-associated bacteria presence

INTERVENTIONS:
Other: In vitro stimulation of blood with periodontitis-associated- and control bacteria — Peripheral mononuclear blood cells are stimulated with periodontitis-associated- and control bacteria to measure the amount of positive cytokine-producing cells.
Diagnostic Test: Anti-CCP- and anti-P.g.-antibodies titers — Anitbody titers will be measured in saliva and serum samples.
Genetic: Analysis of selected single nucleotide polymorphisms (SNPs) — DNA obtained from saliva samples will be used to determine the genotype of the participants for selected SNPs.
Diagnostic Test: periodontitis-associated bacteria presence — Determination of the presence of periodontitis-associated bacteria e.i. Porphyromonas gingivalis in saliva and blood samples.

SUMMARY:
This study evaluates the interaction between host immune cells and bacteria associated with periodontitis. It comprises biological material from donors with and without periodontal disease. Specifically, we collect a spit and blood sample to conduct in vitro stimulations and measurements of selected parameters related to periodontitis to clarify obscure areas in the immunologic pathogenesis of this disease.

DETAILED DESCRIPTION:
Periodontitis is a prevalent, multifactorial inflammatory disease characterized by the interaction between microorganisms organized in biofilms on tooth surfaces and host immune cells, leading to an inflammatory destruction of the tooth-supporting tissues and - if left untreated - eventually tooth loss. Periodontitis affects up to 50% of the population in the United States of America, and is classified in an aggressive and a chronic form depending on genetic factors, age of onset, speed and severity of attachment loss.

The onset of periodontitis is caused by an immunologic imbalance between host immune cells and residing microorganisms in subgingival pockets. The host immune cells are capable of enhancing both a protective and a destructive inflammatory response towards the microorganisms through the release of inflammatory mediators e.i. proinflammatory and antiinflammatory cytokines.

The role of antibodies in periodontitis is also unclear. Some studies show an excessive antibody level against bacteria associated with periodontitis e.g. Porphyromonas gingivalis (P.g.).

In general, this study contributes to a profound understanding of the host immune cells role in the onset and pathogenesis of periodontitis by comparing healthy versus diseased donors immunologic responses toward pathogene and apathogene microorganisms and their genetic background.

ELIGIBILITY:
Inclusion criteria for chronic periodontitis donors:

* 50-60 years of age.
* Interproximal attachment loss at minimum 3 teeth besides molars and incisors.
* Clinical attachment loss at minimum 10 sites identified by bleeding and pus upon probing.
* Visible radiographic bone loss.
* Medically healthy donors.

Inclusion criteria for aggressive periodontitis donors:

* 19-40 years of age.
* Interproximal attachment loss at minimum 3 teeth besides molars and incisors.
* Clinical attachment loss at minimum 10 sites identified by bleeding and pus upon probing.
* Visible radiographic bone loss.
* Medically healthy donors.

Inclusion criteria for healthy donors: (age: 19-40 years; 50-60 years)

* No sign of inflammatory conditions or other general systemic diseases.
* Medically healthy donors.

Exclusion criteria for all groups:

* Pregnant and breastfeeding.
* Antibiotic treatment within 6 months.
* Suffer from periodontal manifestations caused by systemic diseases e.i. genetic diseases, haematologic anomalies or syndromes.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study includes 170 participants, which are legally competent e.i. above 18 years of age and general decision competent. The participants are divided into three groups: 1) Participants with chronic periodontitis (n=35), 2) participants with aggressive periodontitis (n=35) and 3) healthy participants without periodontal disease (n=100). The participants are recruited from the Department of Odontology, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark and assigned to a group in accordance with the periodontal disease classification system in 1999 American Academy of Periodontology.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
periodontitis-associated- and control bacterial stimulation of host immune cells. | Aug. 2020
  Identification and determination of the amount of cytokine-producing immune cells when stimulated with bacteria associated with periodontitis including pro- and antiinflammatory cytokines.
  Genuses: Porphyromonas, Prevotella, Eikenella, Aggregatibacter, Actinomyces, Lactobacillus, Bifidobacterium, Rothia.
Anti-cyclic citrullinated peptides (anti-CCP) antibodies titers. | Aug. 2020
  Determination of the prevalence of anti-CCP-positive periodontitis patients through measure of anti-CCP antibody titers in serum samples and correlation with the level of antibodies to P. gingivalis, and to the abundancy of the bacterium in saliva.
P. gingivalis presence and related antibodies. | Aug. 2020
  Determination of P. gingivalis presence in saliva and serum samples through RT-qPCR and determination of the level of antibodies towards the bacterium using in-house Luminex-based technology.
Single nucleotide polymorphism (SNP) analysis. | Aug. 2020
  Investigation of the potential association between periodontitis and selected polymorphisms in the PADI genes using multiplex bead-based SNP assays with the Luminex technology.

SECONDARY OUTCOMES:
Cytokine profile in saliva. | Aug. 2020
  Determination of the cytokine profile in saliva samples from subject with periodontitis and healthy controls with Luminex based technology.
Presence of other periodontal bacteria. | Aug. 2020
  Determination of the presence of other periodontal bacteria through RT-qPCR assays.

CONTACTS AND LOCATIONS:
Overall Officials: Palle Holmstrup, DDS, PhD, Dr Odont, Study Director — University of Copenhagen; Claus Henrik Nielsen, PhD, MSc, MD, Study Director — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Institute for Inflammation Research, Center for Rheumatology and Spine Diseases, Rigshospitalet, Copenhagen University Hospital., Copenhagen
  - Section for Periodontology, Microbiology and Community Dentistry, Department of Odontology, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers in accordance with our approved Human Subjects Protection application in Denmark.

REFERENCES:
- [Background] Bartold PM, Van Dyke TE. Periodontitis: a host-mediated disruption of microbial homeostasis. Unlearning learned concepts. Periodontol 2000. 2013 Jun;62(1):203-17. doi: 10.1111/j.1600-0757.2012.00450.x. PMID 23574467
- [Background] Neely AL, Holford TR, Loe H, Anerud A, Boysen H. The natural history of periodontal disease in man. Risk factors for progression of attachment loss in individuals receiving no oral health care. J Periodontol. 2001 Aug;72(8):1006-15. doi: 10.1902/jop.2001.72.8.1006. PMID 11525431
- [Background] Eke PI, Dye BA, Wei L, Slade GD, Thornton-Evans GO, Borgnakke WS, Taylor GW, Page RC, Beck JD, Genco RJ. Update on Prevalence of Periodontitis in Adults in the United States: NHANES 2009 to 2012. J Periodontol. 2015 May;86(5):611-22. doi: 10.1902/jop.2015.140520. Epub 2015 Feb 17. PMID 25688694
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Northwest Dent. 2000 Nov-Dec;79(6):31-5. PMID 11413609
- [Background] Haffajee AD, Socransky SS, Patel MR, Song X. Microbial complexes in supragingival plaque. Oral Microbiol Immunol. 2008 Jun;23(3):196-205. doi: 10.1111/j.1399-302X.2007.00411.x. PMID 18402605
- [Background] Damgaard C, Holmstrup P, Van Dyke TE, Nielsen CH. The complement system and its role in the pathogenesis of periodontitis: current concepts. J Periodontal Res. 2015 Jun;50(3):283-93. doi: 10.1111/jre.12209. Epub 2014 Jul 5. PMID 25040158
- [Background] Liu YC, Lerner UH, Teng YT. Cytokine responses against periodontal infection: protective and destructive roles. Periodontol 2000. 2010 Feb;52(1):163-206. doi: 10.1111/j.1600-0757.2009.00321.x. No abstract available. PMID 20017801
- [Background] Kinane DF, Preshaw PM, Loos BG; Working Group 2 of Seventh European Workshop on Periodontology. Host-response: understanding the cellular and molecular mechanisms of host-microbial interactions--consensus of the Seventh European Workshop on Periodontology. J Clin Periodontol. 2011 Mar;38 Suppl 11:44-8. doi: 10.1111/j.1600-051X.2010.01682.x. PMID 21323703
- [Background] Pussinen PJ, Jousilahti P, Alfthan G, Palosuo T, Asikainen S, Salomaa V. Antibodies to periodontal pathogens are associated with coronary heart disease. Arterioscler Thromb Vasc Biol. 2003 Jul 1;23(7):1250-4. doi: 10.1161/01.ATV.0000072969.71452.87. Epub 2003 Apr 24. PMID 12714435
- [Background] Pussinen PJ, Nyyssonen K, Alfthan G, Salonen R, Laukkanen JA, Salonen JT. Serum antibody levels to Actinobacillus actinomycetemcomitans predict the risk for coronary heart disease. Arterioscler Thromb Vasc Biol. 2005 Apr;25(4):833-8. doi: 10.1161/01.ATV.0000157982.69663.59. Epub 2005 Feb 3. PMID 15692101
- [Background] Berglundh T, Donati M. Aspects of adaptive host response in periodontitis. J Clin Periodontol. 2005;32 Suppl 6:87-107. doi: 10.1111/j.1600-051X.2005.00820.x. PMID 16128832
- [Background] Fillatreau S. Cytokine-producing B cells as regulators of pathogenic and protective immune responses. Ann Rheum Dis. 2013 Apr;72 Suppl 2:ii80-4. doi: 10.1136/annrheumdis-2012-202253. Epub 2012 Dec 19. PMID 23253921
- [Background] Belstrom D, Paster BJ, Fiehn NE, Bardow A, Holmstrup P. Salivary bacterial fingerprints of established oral disease revealed by the Human Oral Microbe Identification using Next Generation Sequencing (HOMINGS) technique. J Oral Microbiol. 2016 Jan 14;8:30170. doi: 10.3402/jom.v8.30170. eCollection 2016. PMID 26782357
- [Background] Belstrom D, Holmstrup P, Bardow A, Kokaras A, Fiehn NE, Paster BJ. Comparative analysis of bacterial profiles in unstimulated and stimulated saliva samples. J Oral Microbiol. 2016 Mar 16;8:30112. doi: 10.3402/jom.v8.30112. eCollection 2016. PMID 26987356
- [Derived] Danielsen AK, Damgaard C, Massarenti L, Ostrup P, Riis Hansen P, Holmstrup P, Nielsen CH. B-cell cytokine responses to Porphyromonas gingivalis in patients with periodontitis and healthy controls. J Periodontol. 2023 Aug;94(8):997-1007. doi: 10.1002/JPER.22-0438. Epub 2023 Mar 5. PMID 36715211